CLINICAL TRIAL: NCT02674737
Title: Evaluation of the Effect of Appropriate Sedation for Patients After Gastrectomy: A Prospective Randomised Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Juanhong Shen, Director, PhD, Principal Investigator, Resident Physician, Chinese Medical Association
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jinling37ICUCMH
Record Dates: First submitted 2016-01-21; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Sedation,Gastrectomy, Enhanced Recovery After Surgery
MeSH Terms: interventions — Dexmedetomidine; Tramadol; Flurbiprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine,tramadol and flurbiprofen (Experimental): Both sedative and analgesic(dexmedetomidine, tramadol and flurbiprofen) are applied to this group of patients.
  Interventions: Drug: dexmedetomidine, tramadol and flurbiprofen
- Tramadol and flurbiprofen (Active Comparator): Only routine analgesic(tramadol and flurbiprofen) are applied to this group of patients.
  Interventions: Drug: tramadol and flurbiprofen

INTERVENTIONS:
Drug: dexmedetomidine, tramadol and flurbiprofen
  Arms: Dexmedetomidine,tramadol and flurbiprofen
Drug: tramadol and flurbiprofen
  Arms: Tramadol and flurbiprofen

SUMMARY:
To evaluate the efficacy and safety of appropriate postoperative sedation with dexmedetomidine for patients after gastrectomy. Prospective randomised controlled study was conducted from October 2015 and December 2015 among patients after gastrectomy. The investigators are going to enroll patients who received abdominal surgeries. One group receive sedative along with analgesic and the other group analgesic only for the other group on the first 24 hours after surgeries and follow up for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* underwent gastrectomy in the hospital and operation duration lasted at least 2 hours

Exclusion Criteria:

* take part in other clinical trials
* quinolone antibiotics intake 4 weeks prior to or within the study
* NSAIDS intake within one month
* history of peptic ulcer
* respiratory insufficiency
* renal insufficiency
* acute hepatitis or severe liver disease (Child-Pugh class C)
* pregnancy or lactation
* abnormal ECG with clinical significance
* uncontrolled hypotension
* bleeding tendency or hematological diseases
* untreated mechanical intestinal obstruction
* unable to express or any kind of mental disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain assessed by Prince Henry Pain Scale | 1-3d after gastrectomy
  assessed by Prince Henry Pain Scale by investigators at 8:00 am after surgeries until discharge from ICU
recovery of gastrointestinal function assessed by time to first defecation after surgery | 30 days after gastrectomy
  assessed by time to first defecation after surgery
white blood cell count (10^9/L) | 1-3d after gastrectomy
  evaluate postoperative inflammatory response, blood sample collected at 6:00am for 1-3d after gastrectomy
C-reactive protein (mg/L) | 1-3d after gastrectomy
  evaluate postoperative inflammatory response, blood sample collected at 6:00am for 1-3d after gastrectomy

SECONDARY OUTCOMES:
percentage of time within target sedation range | 1-3d after gastrectomy
  assessed by Richmond Agitation-Sedation Scale by investigators at 8:00 am after surgeries until discharge from ICU, the target range is -2 to +1
risk of bradycardia requiring interventions | 1-3d after gastrectomy
  heart rate <40/min is considered bradycardia
risk of hypotension requiring interventions | 1-3d after gastrectomy
  systolic blood pressure <80 mmHg or/and diastolic blood pressure <50 mmHg is considered hypotension
use of opioids and use of benzodiazepins | 1-3d after gastrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of General Surgery of Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Main results and conclusion will be available